CLINICAL TRIAL: NCT02829762
Title: Precarious Elderly Patient Supported For Cancer Impact on Quality Of Life of a Domotic And Remote Assistance Approach for Elderly Patients Supported For Locally Advanced or Metastatic Cancer, Socially Isolated: Randomized, Comparative, Prospective Multi-Centre Study
Brief Title: Precarious Elderly Patient Supported For Cancer Impact on Quality Of Life of a Domotic And Remote Assistance Approach for Elderly Patients Supported For Locally Advanced or Metastatic Cancer, Socially Isolated
Acronym: PREDOMOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-44; 2015-A01976-43 (Other: ANSM)
Record Dates: First submitted 2016-06-29; First posted 2016-07-12 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Elderly; Locally Advanced or Metastatic Cancer
Keywords: isolated; at risk of isolation; patients
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm PS-DR (Experimental): The interventional arm (PS-DR) will include the implementation of social aids, a monthly social monitoring and home improvement with domotic techniques and remote assistance (in connection with a call center 24h/24).
  Interventions: Other: Program of geriatric and Social intervention associated techniques of Domotic and Remote assistance
- Reference Arm (No Intervention): In the reference arm, patients will have a conventional oncological care, social support measures will be left to the discretion of the clinician and the paramedical team.

INTERVENTIONS:
Other: Program of geriatric and Social intervention associated techniques of Domotic and Remote assistance — Implementation of social aids, a monthly social monitoring and home improvement with domotic techniques and remote assistance
  Arms: Interventional arm PS-DR

SUMMARY:
The objective of the PREDOMOS study is to evaluate the impact of establishing a Program of geriatric and Social intervention associated techniques of Domotic and Remote assistance (PS-DR) on the improvement of quality of life of elderly patients, isolated or at risk of isolation, treated for locally advanced or metastatic cancer.

DETAILED DESCRIPTION:
In France, social isolation and prevalence of cancer increases with the population ageing: it is estimated that in 2050, 1 of 2 cancers will be diagnosed in patients over than 75 years old. Meanwhile, the share of isolated elderly increased from 16 to 24% between 2010 and 2013. It is shown that socially precarious elderly have an increased risk of dying from cancer.

Among the areas of Comprehensive Geriatric Assessment (CGA), social assessment is crucial. It can be assessed by a self-administered 8 items questionnaire, derived from MOS-SS (Medical Outcomes Study Social Support Survey) and validated in the elderly supported for cancer: m-MOS-SS (modified Medical Outcomes Study Social Support).

Once spotted, social isolation can be averted by appropriate measures, provided the intervention of a multidisciplinary team. In this area, the techniques of automation and remote assistance might have an interest. They already demonstrated their impact on falls prevention, addiction, feelings of social isolation and quality of life. However, little is known about the impact of social isolation in elderly patients supported for cancer.

The objective of the PREDOMOS study is to evaluate the impact of establishing a Program of geriatric and Social intervention associated techniques of Domotic and Remote assistance (PS-DR) on the improvement of quality of life of elderly patients, isolated or at risk of isolation, treated for locally advanced or metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* G8 score ≤ 14.
* WHO score ≤2
* Having an ADL score ≥ 4 (Katz scale).
* Having an MMSE score > 24
* At risk of social isolation: m-MOS below 80%, and / or the following criteria: patient living alone without close help (<50 km) and / or primary caregiver of the patient's spouse, spouse limited autonomy and / or reached itself a disease (neurodegenerative disease, cancer disease, other) requiring regular hospital treatment for at least 3 months.
* Locally advanced or metastatic cancer or malignant blood disease (except acute leukemia)
* Treated by chemotherapy, new generation hormone therapy, immunotherapy or targeted therapy in first or second line of treatment, with or without radiotherapy
* Life expectancy more than 6 months
* Informed consent signed.
* Patients affiliated to French social security system in accordance with the French law on biomedical research (Article 1121-11 of the French Code of Public Health)

Exclusion Criteria:

* Patients with other cancers
* Patients should be directed immediately into a rehabilitation and recuperative care service to receive treatment or in a palliative care service
* Inability to sign a consent or under guardianship

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Measure of the quality of life by EORTC-QLQc30 scale 3 months after treatment start | 3 months
  The "global health" score will constitute the main judgment criteria

SECONDARY OUTCOMES:
Time to failure of first line of treatment | From date of inclusion until treatment failure, up to 6 months
  Time between inclusion and treatment failure, whatever the cause
First line of treatment toxicity at the end | 12 months
  Measured by Toxicity scale NCI-CTCAE (National Cancer Institute - Common Terminology Criteria for Adverse Events, version 4.0).
Assessment of the number of chemotherapies received by patient compared to the number of prescribed chemotherapies | 12 months
  Treatment compliance
Assessment of the patient dependency level determined by evaluating the Daily living activities (ADL) with the Katz scale | 3 months and 6 months
Assessment of the patient dependency level determined by evaluating the- instrumental activities across Lawton scale | 3 months and 6 months
Nutritional assessment at 3 months and 6 months | 3 months and 6 months
  Body mass index (BMI) is the ratio of weight to height in cm squared.
Functional assessment at 3 months and 6 months | 3 months and 6 months
  The unipodal station is to stand on one foot without aid. A unipodal station less than 5 seconds indicating a high risk of falls (46).
Overall Survival defined as the time between chemotherapy start and death | up to 12 months
  will be assessed at 6 months and 1 year
Progression free Survival defined as the time between treatment start and the date of first documented progression or death, whatever the cause. | up to 12 months
  Time to progression is the time elapsed between the date of treatment start and the occurrence of progression or relapse if a response was observed (response or stabilization).
  A patient who has not progressed or who did not die at the limit of 1 year will have its censored survival time when tumor enough last evaluation conducted by the deadline of 1 year . The progress will then be defined according to the criteria RECIST1.1 .
  In case of death , it will be identified if it is related to tumor progression , toxicity or complication of treatment or another cause (non-specific death).
Social isolation | 12 months
  Social isolation will be measured by the m -MOS questionnaire. A result < 80% is recognized as the consensus inferior value below which patients are socially isolated position
Measure of the "global health score" to assess the quality of life at first line of treatment | 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Couderc AL, Nouguerede E, Baumstarck K, Loubiere S, Le Caer H, Guillem O, Rousseau F, Greillier L, Norguet-Monnereau E, Cecile M, Boulahssass R, Le Caer F, Tournier S, Butaud C, Guillet P, Nahon S, Kirscher S, Diaz N, Morando C, Villani P, Auquier P, Daumas A. PREDOMOS study, impact of a social intervention program for socially isolated elderly cancer patients: update to the study protocol for a randomized controlled trial. Trials. 2019 Jan 15;20(1):54. doi: 10.1186/s13063-018-3127-0. PMID 30646923
- [Derived] Cretel-Durand E, Nouguerede E, Le Caer H, Rousseau F, Retornaz F, Guillem O, Couderc AL, Greillier L, Norguet E, Cecile M, Boulahssass R, Le Caer F, Tournier S, Butaud C, Guillet P, Nahon S, Poudens L, Kirscher S, Loubiere S, Diaz N, Dhorne J, Auquier P, Baumstarck K. PREDOMOS study, impact of a social intervention program for socially isolated elderly cancer patients: study protocol for a randomized controlled trial. Trials. 2017 Apr 12;18(1):174. doi: 10.1186/s13063-017-1894-7. PMID 28403911